CLINICAL TRIAL: NCT01323894
Title: Osteogenic Effects in Human Mesenchymal Stem Cells Enhanced by Wnt Signaling/Hydroxyapatite Nanoparticles--Comparisons Between Non-viral and Viral Administration in Tissue Engineered Bone Regeneration
Brief Title: Osteogenic Effects in Human Mesenchymal Stem Cells Enhanced by Wnt Signaling
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DMR-99-IRB-122
Record Dates: First submitted 2011-03-24; First posted 2011-03-28 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Primary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The first year purpose:

The best concentration of canonical Wnt3a will be investigated in promoting the osteoblastogenesis of human mesenchymal stem cells.

DETAILED DESCRIPTION:
Our previous work is investigating the viral (Adv-BMP-2) administration for the development of a model to generate bones for possible use in clinical settings; the non-viral and viral administrations will be compared for best osteogenesis effects.

The first year purpose:

The best concentration of canonical Wnt3a will be investigated in promoting the osteoblastogenesis of human mesenchymal stem cells.

ELIGIBILITY:
Inclusion Criteria:

* age above 10 years old
* The patients require surgery ner iliac or abdomen areas

Exclusion Criteria:

* age below 10 years old

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients require surgery ner iliac or abdomen areas
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Osteogenic Effects in Human Mesenchymal Stem Cells Enhanced by Wnt Signaling/Hydroxyapatite Nanoparticles--Comparisons between Non-viral and Viral administration in Tissue Engineered Bone Regeneration | 2 years
  August 2011-July 2013

CONTACTS AND LOCATIONS:
Overall Officials: Sopha Chia-Ning Chang, M.D. Ph.D., Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical Universty Hospital, Taichung, Taiwan